CLINICAL TRIAL: NCT03737812
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Assess the Safety and Efficacy of Elezanumab When Added to Standard of Care in Progressive Forms of Multiple Sclerosis
Brief Title: A Study to Assess the Safety and Efficacy of Elezanumab When Added to Standard of Care in Progressive Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M14-397
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Progressive multiple sclerosis; Elezanumab; ABT-555
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — elezanumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants randomized to receive placebo by intravenous infusion.
  Interventions: Drug: placebo
- Elezanumab 400mg Dose (Experimental): Participants randomized to receive 400mg of elezanumab by intravenous infusion.
  Interventions: Drug: elezanumab
- Elezanumab 1800 mg Dose (Experimental): Participants randomized to receive 1800mg of elezanumab by intravenous infusion.
  Interventions: Drug: elezanumab

INTERVENTIONS:
Drug: elezanumab — solution for infusion
  Other Names: ABT-555
  Arms: Elezanumab 1800 mg Dose; Elezanumab 400mg Dose
Drug: placebo — solution for infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of elezanumab in participants with progressive Multiple Sclerosis (PMS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary-progressive multiple sclerosis (PPMS) or non-relapsing secondary-progressive multiple sclerosis (SPMS) and no relapses for at least 24 months.
* Evidence of physical disability according to Expanded Disability Status Scale (EDSS) or Timed 25-Foot Walk (T25FW) or 9-Hole Peg Test.

Exclusion Criteria:

* Treatment with any of the following within the 6 months prior to Screening: natalizumab; cyclosporine; azathioprine; methotrexate; mycophenolate mofetil; intravenous immunoglobulin (IVIg); any interferon product; and intravenous (IV), oral, or intrathecal corticosteroids for the purposes of disease modification.
* Treatment with the following within 1 year prior to Screening: cyclophosphamide or alemtuzumab.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (30):
  - St. Josephs Hospital and Med Center /ID# 202809, Phoenix, Arizona
  - Sutter East Bay Medical Foundation-Jordon Research and Education Dev. Inst. /ID# 202448, Berkeley, California
  - The Research Center of Southern California /ID# 202802, Carlsbad, California
  - Vladimir Royter MD /ID# 202483, Hanford, California
  - Stanford MS Center /ID# 202445, Palo Alto, California
  - UC Davis Health-Neurological Surgery /ID# 202485, Sacramento, California
  - UCSF School of Medicine - Neurology /ID# 203194, San Francisco, California
  - University of Colorado School of Medicine, Dept of Neurology /ID# 202807, Aurora, Colorado
  - Advanced Neurosciences Research, LLC /ID# 203072, Fort Collins, Colorado
  - Rowe Neurology Institute /ID# 202744, Lenexa, Kansas
  - Duplicate_Parexel International /ID# 202747, Baltimore, Maryland
  - International Neurorehabilitation Institute /ID# 213333, Lutherville, Maryland
  - Michigan Institute for Neurological Disorders (MIND) /ID# 202470, Farmington Hills, Michigan
  - Memorial Neurological Institute and Center for Multiple Sclerosis /ID# 206327, Owosso, Michigan
  - Ridgeview Specialty Clinic Chaska - Neurology /ID# 204384, Chaska, Minnesota
  - Washington University-School of Medicine /ID# 202899, St Louis, Missouri
  - The MS Center for Innovations in Care at Missouri Baptist Medical Center /ID# 205432, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Cent /ID# 204744, Las Vegas, Nevada
  - Oklahoma Med Res. Foundation /ID# 203442, Oklahoma City, Oklahoma
  - Providence Neurological Specialties - West /ID# 203193, Portland, Oregon
  - Advanced Neurosciences Institute /ID# 204555, Franklin, Tennessee
  - KCA Neurology - Franklin /ID# 202912, Franklin, Tennessee
  - Neurology Consultants of Dallas - LBJ Fwy /ID# 203102, Dallas, Texas
  - Central Texas Neurology Consul /ID# 203108, Round Rock, Texas
  - Integrated Neurology Services /ID# 202743, Alexandria, Virginia
  - Evergreen Neuroscience Institute /ID# 204205, Kirkland, Washington
  - Virginia Mason Medical Center /ID# 205439, Seattle, Washington
  - Swedish MS Center /ID# 202904, Seattle, Washington
  - West Virginia Univ School Med /ID# 202849, Morgantown, West Virginia
  - Froedtert Memorial Lutheran Hospital /ID# 202618, Milwaukee, Wisconsin
- Canada (7):
  - University of British Columbia - MS & NMO Clinical Trials Group, Djavad Mowafagh /ID# 203536, Vancouver, British Columbia
  - Duplicate_London Health Sciences Centre - University Hospital /ID# 203538, London, Ontario
  - Ottawa Hospital Research Institute /ID# 203058, Ottawa, Ontario
  - Unity Health Toronto - St. Michael's Hospital /ID# 206213, Toronto, Ontario
  - Recherche Sepmus Inc. /ID# 212852, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CRCHUM /ID# 203869, Montreal, Quebec
  - Montreal Neurological Institut /ID# 203868, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 123 subjects from 35 sites in the United States & Canada were enrolled into the study, were randomized, and received at least 1 dose of study drug. Of these, 108 completed treatment
Period: Overall Study
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose
Started | 43 | 40 | 40
Completed | 38 | 34 | 36
Not Completed | 5 | 6 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Sponsor Discontinued the Study | 4 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — COVID -19 Logistical Restrictions | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose | Total
Number analyzed (Participants) | 43 | 40 | 40 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 39 | 39 | 121
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 14 | 21 | 59
  Male | 19 | 26 | 19 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 3 | 5
  Not Hispanic or Latino | 41 | 40 | 37 | 118
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 42 | 32 | 37 | 111
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 10 | 9 | 32
  United States | 30 | 30 | 31 | 91
Type of MS [Count of Participants; unit: Participants]
  Primary progressive MS (PPMS) | 19 | 21 | 19 | 59
  Non-relapsing secondary progressive multiple sclerosis (nrSPMS) | 24 | 19 | 21 | 64

OUTCOME MEASURES:

1. Primary Outcome: Mean Overall Response Score (ORS)
Description: The ORS is a composite score derived from 4 components: Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), 9-Hole Peg Test in the dominant hand (9HPT-D), and 9HPT in the non-dominant hand (9HPT-ND).
  Clinically significant worsening = -1, no change = 0, clinically significant improvement = +1.
  The ORS is the sum of these scores for the EDSS: Timed 25-Foot Walk, 9-Hole Peg Test-dominant, and 9-Hole Peg Test-nondominant and ranges from -4 to + 4.
Time Frame: Week 52
Population: The Modified Intent-to-Treat (mITT) Analysis Set consists of all randomized subjects who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose
Number analyzed (Participants) | 36 | 31 | 34
score on a scale | -0.74 (0.167) | -0.75 (0.176) | -0.64 (0.170)

2. Secondary Outcome: Disability Improvement Response Rate
Description: Disability improvement response rate is assessed based on the Expanded Disability Status Scale Plus (EDSS+). EDSS+ is comprised of Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW) and 9-Hole Peg Tests (9HPT).
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose
Number analyzed (Participants) | 43 | 40 | 40
Participants | 3 | 7 | 9
Statistical Analysis 1: Comparison: Placebo vs Elezanumab 400mg Dose; Analyzed using a logistic regression model with corresponding baseline value as a covariate and treatment as a main effect. Logistic regression model for EDSS+ includes baseline values for EDSS, Timed 25-Foot Walk, 9-Hole Peg Test-dominant, 9-Hole Peg Test-nondominant, and treatment as a main effect. Subjects with missing values were imputed as non-responders; Test type: Other — a statistical test was not performed; Odds Ratio (OR) = 2.230, 95% CI 2-sided [0.485 to 10.259]
Statistical Analysis 2: Comparison: Placebo vs Elezanumab 1800 mg Dose; [analysis description as in outcome 2, analysis 1]; Test type: Other — a statistical test was not performed; Odds Ratio (OR) = 3.859, 95% CI 2-sided [0.899 to 16.561]

3. Secondary Outcome: Overall Response Score (ORS)
Description: The ORS is a composite score derived from 4 components: Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), 9-Hole Peg Test in the dominant hand (9HPT-D), and 9HPT in the non-dominant hand (9HPT-ND).
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose
Number analyzed (Participants) | 38 | 35 | 34
score on a scale | -0.47 (0.134) | 0.00 (0.136) | -0.21 (0.139)

4. Secondary Outcome: Overall Response Score (ORS)
Description: The ORS is a composite score derived from 4 components: Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), 9-Hole Peg Test in the dominant hand (9HPT-D), and 9HPT in the non-dominant hand (9HPT-ND).
  Clinically significant worsening = -1, no change = 0, clinically significant improvement = +1.
  The ORS is the sum of these scores for the EDSS, Timed 25-Foot Walk, 9-Hole Peg Test-dominant and 9-Hole Peg Test-non-dominant and ranges from -4 to + 4.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose
Number analyzed (Participants) | 36 | 28 | 31
score on a scale | -0.28 (0.176) | -0.27 (0.194) | -0.53 (0.188)

5. Secondary Outcome: Overall Response Score (ORS)
Description: as for outcome 4
Time Frame: Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose
Number analyzed (Participants) | 35 | 26 | 30
score on a scale | -0.45 (0.159) | -0.48 (0.178) | -0.52 (0.169)

ADVERSE EVENTS:
Time Frame: Up to 76 weeks
Description: Adverse Events were collected for all study participants, whether solicited or spontaneously reported by the study participant throughout the study, who received at least 1 dose of study drug and for a period of up to 39 weeks after the last dose of study drug.
Arm/Group | Placebo | Elezanumab 400mg Dose | Elezanumab 1800 mg Dose
All-Cause Mortality (participants affected / at risk) | 1/43 | 1/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/43 | 5/40 | 3/40
Other Adverse Events (participants affected / at risk) | 34/43 | 29/40 | 31/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Elezanumab 400mg Dose (N=40) | Elezanumab 1800 mg Dose (N=40)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
UHTHOFF'S PHENOMENON (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Elezanumab 400mg Dose (N=40) | Elezanumab 1800 mg Dose (N=40)
VERTIGO (Ear and labyrinth disorders) | 3 (4) | 3 (3) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (14) | 2 (2) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
CHEST DISCOMFORT (General disorders) | 0 (0) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 4 (6) | 6 (7) | 6 (6)
PAIN (General disorders) | 0 (0) | 2 (2) | 3 (3)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (2)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (3) | 3 (7)
URINARY TRACT INFECTION (Infections and infestations) | 7 (14) | 8 (9) | 9 (10)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 6 (13) | 4 (4) | 9 (15)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 5 (8) | 2 (4) | 8 (13)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (5) | 2 (3)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (3)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1)
DIZZINESS (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 7 (20) | 5 (9) | 4 (5)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
MUSCLE SPASTICITY (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
NEURALGIA (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 2 (2) | 2 (3)
DEPRESSION (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
INSOMNIA (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (2)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT03737812/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03737812/SAP_001.pdf